CLINICAL TRIAL: NCT05431140
Title: Evaluation of CloudCare in the Treatment of Type 1 Diabetes. A Prospective Cohort Study in the Netherlands
Brief Title: Evaluation of CloudCare in the Treatment of Type 1 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Diabeter Nederland BV (Other)
Responsible Party: Sponsor
Other Study IDs: DIA-2022-01
Record Dates: First submitted 2022-06-21; First posted 2022-06-24 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Type 1 Diabetes
Keywords: cohort; prospective; observational
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CloudCare — Only eligible subjects to whom CloudCare is introduced as part of their new standard care will be enrolled. Participants will not be subjected to extra procedures on top of their standard of care, except that they will be asked to fill out short questionnaires about their treatment satisfaction and the emotional burden caused by diabetes, which are not standard in the participating study locations.

SUMMARY:
CloudCare is an eHealth application to help health care professionals (HCP) in the management/treatment of type 1 diabetes. The application will automatically check all uploaded glucose parameters from patients glucose monitoring devices and present all these data in a categorized way (using a so called dashboard) to the HCP. In this way the HCP has a direct overview of the condition of her/his patients, and can determine which data request direct action towards the patient and which data do not. It is expected that this system improves outcome and patient experience.

In this study this expectation will be studied by measuring the effect of CloudCare on patients' treatment satisfaction, glucose control, HCP satisfaction and the impact on costs.

DETAILED DESCRIPTION:
Diabeter offers a Conformité Européenne (CE) marked eHealth application called CloudCare. This is a customizable care management and decision support system that uses algorithms and automation to help triage clinically relevant cases from all incoming data transmission (data uploads) and improve clinical workflows. This should complement existing clinical care models, like face-to-face meetings. The CloudCare application offers the Health Care Professional (HCP) a better and accurate oversight of the patient's condition, which enables the HCP to contact the patient in a timely manner. CloudCare enables improved use of clinically relevant data by both patients and care team and is expected to improve outcomes and patient experience.

This prospective cohort study aims to estimate the effect of the CloudCare application in daily practice on patients' treatment satisfaction, glycaemic control ('glucometric'), HCP satisfaction and the impact on costs.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign the study informed consent form prior to any data collection for this study
* Clinical diagnosis, based on investigator assessment, of type 1 diabetes and using insulin with or without metformin for at least 6 months.
* Age between 16 and 75 years old.
* Use of multiple daily injections of insulin (MDI, with a basal insulin injection and bolus injections) or continuous subcutaneous insulin infusion (CSII) with Flash or Continuous Glucose Monitoring (FGM/CGM), but without CloudCare for at least three months.
* Receiving CloudCare as part of their standard care for at least 6 months.

Exclusion Criteria:

* Patients with type 1 diabetes on glucose lowering treatments other than insulin with or without metformin.
* Any known factor, condition, or disease that might interfere with study conduct or interpretation of the results, as deemed by the investigator.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 194 adult patients with type 1 diabetes (16-75 years) will be enrolled into the study. All participants must be treated with multiple daily injections of insulin (MDI) or continuous subcutaneous insulin infusion (CSII) with continuous or flash glucose monitoring (CGM/FGM) for at least three months without CloudCare and will get CloudCare as part of their standard care.
Sampling Method: Non-Probability Sample
Enrollment: 194 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Diabetes Treatment Satisfaction Questionnaire (DTSQc) | after 3 and 6 months
  Change in mean patient treatment satisfaction score at 3 and 6 months (prospective) using change version of the DTSQc

SECONDARY OUTCOMES:
% HbA1c | -3 (postspective) , +3 and +6 months (prospective)
  Change in mean % HbA1c at 3 and 6 months
Time in Range (TIR) | -3 (postspective) , +3 and +6 months (prospective)
  Change in mean TIR at 3 and 6 months
Time above Range (TAR) | -3 (postspective) , +3 and +6 months (prospective)
  Change in mean TAR at 3 and 6 months
Time below Range (TBR) | -3 (postspective) , +3 and +6 months (prospective)
  Change in mean TBR at 3 and 6 months
Problem Areas In Diabetes (PAID-5) questionnaire score | after 3 and 6 months
  Change in mean PAID-5 questionnaire score
Change in mean treatment satisfaction score of the HCP satisfaction Questionnaire | after 3 and 6 months
  Self developed questionnaire. Not validated
Number of reported complications requiring hospitalizations | -3 (postspective) , +3 and +6 months (prospective)
  Number of Serious Adverse Events (SAEs) that fulfill the definition of hospitalization
Treatment costs of complications requiring hospitalizations | -3 (postspective) , +3 and +6 months (prospective)
  Costs for hospitalization
Number of contacts with HCP | -3 (postspective) , +3 and +6 months (prospective)
  Number of contacts of patient with HCP during 3 months time period
Type of contacts with HCP | -3 (postspective) , +3 and +6 months (prospective)
  Face to face, Email/Telephone
Time spent by the HCP | -3 (postspective) , +3 and +6 months (prospective)

CONTACTS AND LOCATIONS:
Overall Officials: Henk-Jan Aanstoot, MD, Principal Investigator — Diabeter Nederland B.V.
Locations (1):
- Diabeter, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van Beers CAJ, Last S, Dekker P, Birnie E, Riegman N, van der Pluijm F, Fransman C, Veeze HJ, Aanstoot HJ. Evaluating cloudcare, a population health management system, in persons with type 1 diabetes: an observational study. BMC Endocr Disord. 2025 Mar 31;25(1):88. doi: 10.1186/s12902-025-01905-4. PMID 40165180